CLINICAL TRIAL: NCT01464008
Title: The Predictive Values of Rapid Virus Response and Complete Early Virus Response for Sustained Virus Response in Chronic Hepatitis C Treated With Individual Therapeutic Programme
Brief Title: The Predictive Value of On-treatment Virological Response for Sustained Virological Response in Chronic Hepatitis C
Status: Completed | Type: Observational
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Yao Xie, Head of liver diseases center, Beijing Ditan Hospital
Other Study IDs: DTH-XY001
Record Dates: First submitted 2011-10-28; First posted 2011-11-02 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- chronic hepatitis C
  Interventions: Drug: Pegylated interferon alfa-2a and ribavirin

INTERVENTIONS:
Drug: Pegylated interferon alfa-2a and ribavirin — all patients were given peginterferon alfa-2a (40KD) (Pegasys®; Roche, Basel, Switzerland) 135 or 180 µg by subcutaneous injection once weekly, and received twice daily oral ribavirin at a target total daily dose of 13 mg/kg/day. .
  Other Names: Pegasys®; Roche, Basel, Switzerland

SUMMARY:
The efficacy of combination antiviral therapy for chronic hepatitis C is influenced by many factors. Important patient-specific factors include, age, gender, race, body weight. Important virus-specific factors include HCV genotype and serum HCV RNA level. Finally, important treatment-related factors include the type of interferon, dose of ribavirin and the duration and adherence to treatment.

Despite the importance of patient- and virus-specific factors, the most important indicator of treatment success is a rapid, profound and sustained decrease in serum HCV RNA levels after the start of treatment.

The on-treatment virological response can thus be used to predict the probability that a given patient will achieve an SVR if they remain on therapy. It can also be used to individualize the duration of treatment.

In this study, treatment for patients with chronic hepatitis C was individualized on the basis of clinical characteristics and the on-treatment virological response. The aim was to investigate the usefulness of undetectable HCV RNA levels at week 4 (RVR) and 12 in tailoring the duration of treatment and predicting SVR in Chinese patients with chronic hepatitis C.

DETAILED DESCRIPTION:
297 consecutive patients with chronic hepatitis C who were admitted to hospital or treated as outpatients at Beijing Ditan Hospital were eligible for the study. The diagnosis of chronic hepatitis C was based on the detection of anti-HCV antibodies (anti-HCV) by a third generation microparticle chemoluminescence assay and HCV RNA by a reverse transcription polymerase chain reaction (RT-PCR) assay. Patients were required to have evidence of HCV infection for at least 6 months.

patients received peginterferon alfa-2a (40KD) (Pegasys®; Roche, Basel, Switzerland) 135 or 180 µg by subcutaneous injection once weekly.

Among treatment-naive patients, the duration of therapy was determined by HCV genotype and the on-treatment virological response at week 4, 12 or 24. Genotype 1 infected patients were assigned to complete a 48~72 weeks of treatment, and those who had not responded to a previous course of therapy were assigned to complete a total of 72 weeks of treatment.

Dose adjustment: In the event that a patient did not achieve an RVR at week 4, and provided they were not experiencing adverse events, the daily dosage of ribavirin was increased by 200 mg or 300 mg, and in the case of those who started treatment on the lower dosage of peginterferon alfa-2a (40KD) or conventional interferon alfa, the dosage of peginterferon alfa-2a (40KD) was increased from 135 µg/week to 180 µg/week. In the event of adverse events that could not be ameliorated with symptomatic treatment, the dose of peginterferon alfa-2a (40KD) was reduced from 180 µg/week to 135 µg/week and of ribavirin by 200 mg/day or 300 mg/day.

Quantitative HCV RNA testing was performed before starting treatment (week 0), at week 4, 12, and 24, and at the end of treatment, and 24 weeks after completion of treatment using a commercially available real-time fluorescence quantitative PCR kit. The primary efficacy end-point was achievement of SVR defined as undetectable HCV RNA at the end of a 24-week untreated follow-up period. The percentage of patients with undetectable HCV RNA (<500 copies/mL) at week 4 (RVR), and 12 were secondary efficacy endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Patients with anti-HCV and HCV RNA positive for at least 6 months

Exclusion Criteria:

* Had a haemoglobin level <100 g/L
* Neutrophil count <1.5 x 109/L
* Platelet count <50 x 109/L
* Decompensated liver cirrhosis or liver disease other than that attributable to chronic hepatitis C
* Co-infected with hepatitis B virus or human immunodeficiency virus
* Had an autoimmune disease, liver tumour, or severe cardiac disease.

Ages: 11 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients with chronic hepatitis C who were admitted to hospital or treated as outpatients at Beijing Ditan Hospital were eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 297 (Actual)
Dates: Start 2004-01; Primary Completion 2011-05 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Sustained virus response | serum HCV RNA was undetectabale at the end of treatment and 24 weeks follow
  after treatment, the HCV RNA levels were tested before treatment, at week 4, 12, and 24, and at the end of treatment, and 24 weeks after completion of treatment. The sustained virus response was defined as HCV RNA undetectabale at 24 week after completion of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yao Xie, phD/MD, Study Director — Beijing Ditan Hospital
Locations (1):
- Beijing Ditan hospital,Capital Medical University, Beijing, Beijing Municipality, China